CLINICAL TRIAL: NCT00759005
Title: Effect of Stress on Heroin-Related Memory Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Dependence, China (Other)
Other Study IDs: NIDD
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Heroin Dependence; Learning and Memory
MeSH Terms: conditions — Heroin Dependence | interventions — Propranolol; Hydrocortisone

ARMS (1):
- A, 4 (Experimental)
  Interventions: Drug: propranolol and cortisol

INTERVENTIONS:
Drug: propranolol and cortisol

SUMMARY:
The purpose of this study is to determine whether cortisol and propranolol are effective in the modulation of stress induced heroin-related retrieval enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Participants had to have met DSM-IV criteria for heroin dependence prior to abstinence.

Exclusion Criteria:

* current use of any medications; current DSM-IV diagnosis of any affective, anxiety, or psychotic disorder; current dependence on any substance besides heroin and nicotine (based on DSM-IV criteria); or risk factors for untoward side effects from propranolol and cortisol (i.e., irregular heartbeats, history of cardiogenic shock, history of severe heart failure, asthma, fungal Infections, hyperlipidemia, history of hypertension, or abnormal ECG or other laboratory findings).

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Glucocorticoids enhanced heroin-related memory retrieval in abstained heroin addicts

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Dependence, Beijing, Beijing Municipality, China